CLINICAL TRIAL: NCT02313259
Title: The Impact of Ocular Diseases on Driving: a Prospective Study
Status: Completed | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-1593, DR-002-1370
Record Dates: First submitted 2014-08-25; First posted 2014-12-10 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2015-09

CONDITIONS: Macular Degeneration; Glaucoma
MeSH Terms: conditions — Macular Degeneration; Glaucoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- AMD controls: 15 patients with early to intermediate AMD (grade 2-8) were enrolled using the Age-Related Eye Disease Study (AREDS) severity scale for AMD.
  Interventions: Other: Speed discrimination test; Behavioral: Driving simulation
- Age-matched controls: 15 drivers without ocular disease.
  Interventions: Other: Speed discrimination test; Behavioral: Driving simulation
- Young controls: 15 drivers without ocular disease. Between 18 and 25 years old.
  Interventions: Other: Speed discrimination test; Behavioral: Driving simulation
- Glaucoma patients: 15 patients having a Humphrey visual field mean deviation between -10 and -12 (better eye).
  Interventions: Behavioral: Driving simulation

INTERVENTIONS:
Other: Speed discrimination test — The participant has to stare in the middle of two screens, i.e the reference screen and the test screen. Dots are moving from the center to the edge of the screens at different speeds. The participant is forced to determine if the dots of the test screen are moving faster or slower than the reference screen.
  The test is designed in Psychtoolbox3. Data analyses performed using MATLAB. Two-alternative forced choice paradigm.
  Groups: AMD controls; Age-matched controls; Young controls
Behavioral: Driving simulation — 25 km simulated car driving session. The participant is seated in the driver compartment of a real car featuring all the actual components (steering wheel, pedals regulating speed and brakes). He is instructed to respect road regulations as well as safety rules and must perform some driving manoeuvres, such has turning at intersections, stopping when necessary, passing another car, etc.
  Software Drive 3.0 by Systems Technology Inc., Hawthorne, California, USA. Magnetic head tracker (Flock of Birds, Ascension Technology Corporation, Burlington, Vermont, USA).
  A fixed-base driving simulator. 2 driving scenarios: a practice (10 minutes) and a main scenario including rural and urban sections (35 minutes).

SUMMARY:
The purpose of the study was (1) to determine thresholds for discriminating speed in peripheral fields of patients with dry AMD and (2) to examine the driving skills of licensed drivers with early dry AMD using a driving simulator and to investigate how their healthy counterparts perform on the same driving tasks. We hypothesized that speed discrimination may be better in patients with dry AMD than in healthy control subjects.

DETAILED DESCRIPTION:
This observational study has two goals:

1. to establish if patients affected by dry AMD have a different speed discriminating threshold using peripheral vision fields than their healthy counterparts.
2. to determine if the driving skills of AMD and glaucoma patients differ from healthy controls.

Two tasks will be used: 1) A speed discrimination test. (Glaucoma patient are not asked to perform this task as it assesses the peripheral visual fields, which is affected by the disease.) 2) A driving simulation session. Participant will undergo both tests on the same day, no later than a month after the initial recruitement visit.

For both diseases, patients will be compared to healthy controls matched for age and gender, but also to a younger control group. The latter group was added in order to take into account the normal aging impact on driving skills (visual and cognitive).

Our hypothesis is that AMD patient will show a better speed discriminating threshold than matched control and maybe better or equal to the younger control groups. We also hypothesize that driving skills involving peripheric speed awareness, such as passing another car, will be enhanced in the AMD group when compared to glaucoma patients and age-matched control group.

ELIGIBILITY:
Inclusion Criteria:

* Best-corrected visual acuity (BCVA) had to be at least 20/50 (6/15).
* Binocular visual field (VF) should not be less than 120° along the horizontal meridian and 20° above and below the same meridian.
* Valid driving license
* Diagnosis of bilateral dry AMD (AMD group) or open-angle glaucoma (glaucoma group)

Exclusion Criteria:

* Diplopia
* Cognitive impairment
* Other ocular diseases

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients (with glaucoma or AMD) were recruited from the Centre Universitaire d'Ophtalmologie (CUO), Saint-Sacrement Hospital in Quebec City.
  Participants in control groups are residents of Quebec City.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2015-02-23 (Actual); Study Completion 2015-02-23 (Actual)

PRIMARY OUTCOMES:
Speed discrimination threshold | Before driving simulation
  75% point is taken as a measure of the discrimination threshold.

SECONDARY OUTCOMES:
Driving performance | After speed discrimination task
  Probe reaction time task. Speed limits. Respect of traffic safety rules.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Lalonde, MD, Principal Investigator — Centre Universitaire d'Ophtalmologie (CUO), Saint-Sacrement Hospital, Quebec City.; Marc Hébert, PhD, Study Director — Centre Universitaire d'Ophtalmologie (CUO), Saint-Sacrement Hospital, Quebec City
Locations (1):
- Centre universitaire d'ophtalmologie, Hôpital du Saint-Sacrement, CHU de Québec, Québec, Quebec, Canada